CLINICAL TRIAL: NCT04778280
Title: Estimation of Vitamin D in Humans Infected With Giardia Lamblia
Brief Title: Vitamin D Estimation With Giardia Lamblia Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Sayed Farrag, principlal investigator, Sohag University
Other Study IDs: Soh-Med-21-02-17
Record Dates: First submitted 2021-02-25; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Giardia Lamblia Infection
Keywords: estimaion of vitamin D in humans infected with Giardia lamblia
MeSH Terms: conditions — Giardiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: 1-Group A(Healty group with negative Giardia lamblia or control group) 96 samples
- Group B: 2- Group B(Cases group with positive Giardia lamblia )96 sample

SUMMARY:
investigators will take stool and blood samples from two groups of humans :-

1-group A (healthy group negative Giardia or control group),2-group B (positive Giardia or case group)then investigators make estimation for vitamin D in both groups then investigators try to find if there is relation between vitamin D level and Giardia lamblia infections

DETAILED DESCRIPTION:
In this research a case- control study will be used) ,the percentage of case to control will be 1:1 the total number of samples 192 ,investigators will take stool and blood samples from two groups of humans :-

1-group A (healthy group negative Giardia or control group),2-group B (positive Giardia or case group)then investigators make estimation for vitamin D in both groups then investigators try to find if there is relation between vitamin D level and Giardia lamblia infections

ELIGIBILITY:
Inclusion Criteria:

* patient infected with Giardia lamblia.

Exclusion Criteria:

* patient takes vitamin D supplement - patient has kidney disease- patient has liver disease-patient has a debilitating disease disease such as cancer or diabetes.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: we take 192 samples then we will divide these samples into two groups :-
  1. Group A (healty group with negative Giardia lamblia or control group)
  2. Group B ( diseased group with positive Giardia lamblia or cases group)
Sampling Method: Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
fluctuation level of vitamin D level | 1 year
  Estimation of vitamin D level in humans infected with Giardia lamblia

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Sayed Farrag, Demonstrator, Principal Investigator — faculty of medicine sohag university; Mohammed Sayed Farrag, Demonstrator, Study Director — faculty of medicine sohag university
Locations (2):
- Egypt (2):
  - Faculty of Medicine Sohag University, Sohag
  - Faculty of Medicine, Sohag